CLINICAL TRIAL: NCT02639715
Title: Morphometrics and Morphokinetics of Thawed Oocytes and Embryos
Status: Completed | Type: Observational
Sponsor: Sophie Debrock (Other)
Responsible Party: Sponsor-Investigator, Sophie Debrock, Professor Doctor PhD, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S55685
Record Dates: First submitted 2015-12-15; First posted 2015-12-24 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this observational study is to describe for the first time a complete set of morphometric and morphokinetic parameters of frozen-thawed human embryos in order to select the embryo with the highest implantation potential. These parameters will be correlated with (1) data of the fresh embryos and their subsequent survival, the evolution of the contact surfaces between surviving blastomeres and the resumption of mitosis; (2) patient characteristics and clinical outcome of frozen-thawed embryos and (3) a comparison between embryos cryopreserved with vitrification or the slow method regarding these parameters will be performed.

This project aims to introduce new evaluation criteria of the frozen-thawed embryos to improve success rate of FET cycles. By establishing new precise, reliable and non-invasive measurable parameters, we aim to (1) select which supernumerary embryos are at chance to survive the freezing/thawing procedures, (2) establish cut off parameters for the survival rate of the embryo, (3) assess implantation, pregnancy and live birth rates depending on the developmental characteristics after thawing and after 24h of culture.

Our strategy for improving the outcome of FET cycles is based on the study of morphometric and morphokinetic parameters in frozen-thawed embryos and the correlation with embryological, clinical and cycle parameters. Transferring a well-defined thawed embryo with a high implantation potential may lead towards an increase in the implantation and life birth rate and an increase in the cumulative live birth rate with a reduction of the IVF costs in order to optimize the health-economic situation of reproductive medicine.

DETAILED DESCRIPTION:
Cryopreservation of supernumerary embryos is an essential part of Assisted Reproduction Techniques (ART) and is nowadays a standard routine procedure in the IVF laboratory. Its clinical application consists in (1) the possibility of increasing cumulative delivery rates per cycle and (2) the reduction of the number of transferable embryos in both fresh and successive frozen thawed embryo transfer cycles (FET) decreasing the risk of multiple pregnancies.

Two different techniques to cryopreserve embryos are commonly used: slow freezing and vitrification. During slow freezing, the embryo is exposed to subzero temperatures in a controlled rate with the use of low concentration of cryoprotectant. Alternatively, using vitrification the embryo rapidly enters into a glass-like state with the use of high concentrations of cryoprotectant and rapid cooling rates. Several studies comparing cryopreservation of human embryos by vitrification or slow freezing are available and meta-analyses have been published. Although vitrification has been found to have significantly higher survival rates than slow freezing, results on implantation rate, clinical pregnancy rate and live birth rate remain unclear, mostly due to a paucity of well-designed and powered prospective randomized controlled studies assessing live birth rates.

Embryo evaluation to select the embryo(s) with the highest implantation potential is routinely based on embryo developmental and morphological characteristics using light microscopy. The embryo parameters usually correlated to the implantation capacity of an embryo in a fresh cycle are the number of blastomeres, their symmetry and the percentage cytoplasmic fragmentation. For the evaluation of frozen-thawed embryos, the percentage of blastomeres that survive the freezing-thawing process and their developmental capacity after overnight culture have to be added to these factors.

Current research in the development of non-invasive methods for scoring embryos and ranking them according to their ability to implant and give rise to a healthy birth include both morphometrics and morphokinetics.

Morphometrics Multilevel computerized images enable assessment over an unlimited time period and allow a detailed evaluation of the embryo. Several morphometric studies of human fresh oocytes and embryos with embryo implantation and development have been published. Morphometric studies using multilevel images combined with a computer-assisted scoring system (CASS) may be superior compared to standard scoring system (SSS) to predict implantation and/or live birth based on the number and size of blastomeres on day 3. Semi-automated morphometric analysis also revealed correlations between total embryo volume and clinical pregnancy. Another study evaluating morphometric characteristics including the absolute volumes, coefficients of form and the coefficient of diversity of human embryos and/or oocytes showed a higher coefficient of diversity between sister blastomeres in embryos that successfully implanted and progressed to birth. Morphometric characteristics including the external and internal diameter of the zona pellucida, the thickness of the zona pellucida and the embryo cell mass diameter were described. They stated that image analysis could be used to predict the criteria needed for more efficient embryo assessment before transfer. The mean blastomere size was correlated with the degree of fragmentation and multinucleation in a study using computer-controlled multilevel analyses with 232 embryos. However, until now, no morphometric studies in human frozen thawed embryos have been described.

Morphokinetics Time-lapse imaging allows documentation of early growth without disturbing the culture environment. At this moment, no prospective randomized trial data are available showing that embryos selected from time-lapse imaging have significantly improved implantation rates compared with embryos selected with conventional morphological evaluation.

However, time lapse imaging of embryos have revealed a correlation between first cleavage time, time between cleavages, blastomere size and multinucleation and implantation potential of human embryos. A correlation between the times of each embryo cleavage between 2 to 8 cell stage, the ability to become a blastocyst and implantation potential. Moreover, morphokinetic studies have demonstrated that direct cleavage from 2 cells to 3 cells has been correlated with a low implantation and ongoing pregnancy rate. According to time-lapse recording in 38 oocytes, embryo quality was related to fertilization events and periodicity of the cyctoplasmic wave: good quality embryos arose from oocytes that had more uniform timing from injection to pronuclear abuttal and longer cytoplasmic wave. Furthermore, cellular fragments in human embryos can disappear during in vitro culture.

Only a few studies on morphokinetics in human cryopreserved embryos have been published. Using videocinematography on respectively 50 and 103 frozen-thawed embryos, it was shown that the occurrence of smooth membranes and the cell-cell adherence were predictive for the implantation capacity of frozen-cleaved embryos. Wong et al. followed the development of 242 supernumerary frozen d1-old embryos in a study combining time lapse microscopy and gene expression profiling: success in progression to the blastocyst stage could be predicted by measuring three dynamic, noninvasive imaging parameters by day 2 after fertilization before embryonic genome activation: (1) duration of the first cytokinesis, (2) time interval between the end of the first mitosis and the initiation of the second and (3) the time interval between the second and third mitoses.

This observational study aims to describe morphometric and morphokinetic parameters of thawed human embryos after freezing (slow freezing or vitrification). The study will focus on the evolution of the blastomere volume, the evolution of the contact surfaces between surviving blastomeres and the development of the embryo using time lapse imaging. Embryo morphometric and morphokinetic parameters will be analyzed together with patient characteristics and clinical parameters using cluster analysis techniques. The correlation between morphometrics/morphokinetics and the implantation potential of frozen-thawed embryos will be studied in cycles with single embryo transfer and in cycles with dual implantation after double embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* patients with female age < 40 years at Oocyte retrieval

Exclusion Criteria:

* Patients with female age >40 years at Oocyte retrieval
* cycles with Preimplantation genetic diagnosis
* donated gametes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with frozen thawed embryos for an ART treatment cycle
Sampling Method: Non-Probability Sample
Enrollment: 1272 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
embryo implantation (measured by the number of intrauterine fetal sacs on ultrasound per number of embryos transferred) after a thawing / warming cycle | 6-7 weeks

REFERENCES:
- [Derived] Fernandez Gallardo E, Spiessens C, D'Hooghe T, Debrock S. Effect of day 3 embryo morphometrics and morphokinetics on survival and implantation after slow freezing-thawing and after vitrification-warming: a retrospective cohort study. Reprod Biol Endocrinol. 2017 Oct 3;15(1):79. doi: 10.1186/s12958-017-0299-5. PMID 28974230
- [Derived] Fernandez Gallardo E, Spiessens C, D'Hooghe T, Debrock S. Effect of embryo morphology and morphometrics on implantation of vitrified day 3 embryos after warming: a retrospective cohort study. Reprod Biol Endocrinol. 2016 Jul 30;14(1):40. doi: 10.1186/s12958-016-0175-8. PMID 27475526